CLINICAL TRIAL: NCT03264326
Title: Efficacy of Blood Flow Restriction Training Combined With Eccentric Exercise as Assessed by Shear Wave Elastography in Subjects With Chronic Achilles Tendinopathy: A Randomized Single Blinded Controlled Trial
Brief Title: Efficacy of BFR Training Combined With Eccentric Exercise as Assessed by SWE in Subjects With Chronic AT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left institution and not enough resources to support at MTF
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other); Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161202
Record Dates: First submitted 2017-08-02; First posted 2017-08-29 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant blinded to group assignment, assessor blinded to group assignment, investigator blinded to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR Group (Experimental): Blood Flow Restriction Training with Eccentric Exercise Protocol
  Interventions: Other: Blood Flow Restriction Training; Other: Eccentric Exercise
- Sham BFR Group (Sham Comparator): Sham Blood Flow Restriction Training with Eccentric Exercise Protocol
  Interventions: Other: Sham Blood Flow Restriction Training; Other: Eccentric Exercise

INTERVENTIONS:
Other: Blood Flow Restriction Training — Delfi Personalized Tourniquet System occludes 80% venous pressure during lower extremity exercise.
  Arms: BFR Group
Other: Sham Blood Flow Restriction Training — Delfi Personalized Tourniquet System occlude 20 mmHG venous pressure during lower extremity exercise as a sham treatment.
  Arms: Sham BFR Group
Other: Eccentric Exercise — Subjects perform eccentric calf lowering off a step for 90 repetitions twice daily.

SUMMARY:
The purpose of this randomized controlled trial is to use Shear Wave Elastography (SWE) to assess Achilles tendinopathy and the effectiveness of Blood Flow Restriction (BFR) training in patients with Achilles tendinopathy as measured by Numeric Pain Rating Scale, functional self-report, and objective functional measures. SWE will be utilized to objectively quantify tendon properties and BFR training and eccentric exercise will be utilized to treat Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Achilles pain for > 3 months
* Unilateral symptoms only
* DOD beneficiary, between the ages of 18 and 65
* Clinical diagnosis of Achilles tendinopathy
* Read and speak English well enough to provide informed consent and follow study instructions.
* Can attend in-clinic treatments 2-3 x weekly for the next 12 weeks

Exclusion Criteria:

* Any disease or disease process that would preclude the participant from safely performing any of the exercises or intervention at the discretion of the PI. (Uncontrolled diabetes, cardiac disease, severe COPD, open wounds, current infection, etc.)
* Any LE surgery on either side in the last 2 years
* History of Achilles rupture
* Any vascular disorder (varicose veins, Hx of DVT)
* Leaving post/station in the following 3 months precluding them being able to come in for f/u visits
* Self-report of pregnancy (currently or within last 6 months)
* Other foot/LE disorder that prevents the completion of the eccentric exercises or BFR exercise
* Unable/unwilling to hop on symptomatic leg
* Pain < 2/10 of average pain on NPRS
* VISA A score > 80%
* Currently going through MEB/worker's comp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Shear Wave Elastography velocity | At baseline.
  Difference between involved and uninvolved Achilles tendon
VISA-A | From baseline to 24 weeks
  Change in subjective self-report of Achilles function

SECONDARY OUTCOMES:
Triple hop test | At baseline, then at 3 weeks, 6 weeks, 9 weeks, and 12 weeks.
  Distance in length of 3 consecutive hops on one foot
SL Calf Raise Endurance | At baseline, then at 3 weeks, 6 weeks, 9 weeks, and 12 weeks.
  Number of single leg calf raises to failure
SL Jump Height | At baseline, then at 3 weeks, 6 weeks, 9 weeks, and 12 weeks.
  Distance in height of single leg jump
Thigh Circumference | At baseline, then at 3 weeks, 6 weeks, 9 weeks, and 12 weeks.
  circumferential measurement of thigh
Calf Circumference | At baseline, then at 3 weeks, 6 weeks, 9 weeks, and 12 weeks.
  circumferential measurement of calf
Numerical Pain Rating Scale | At baseline, then at 3 weeks, 6 weeks, 9 weeks, 12 weeks and 24 weeks.
  Pain level on a 0 to 10 scale
Global Rating of Change | At 3 weeks, 6 weeks, 9 weeks, 12 weeks and 24 weeks.
  15 point Likert scale from -7 to +7
Shear Wave Elastography velocity | Baseline, at 3 weeks, 6 weeks, 9 weeks, 12 weeks.
  Change in shear wave elastography of symptomatic Achilles tendon over time.

OTHER OUTCOMES:
Blinding/Group assignment assessment | At 12 weeks and 24 weeks.
  Question asking which group they believe they are in (interventional vs control)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Whitehurst, DPT, Principal Investigator — Womack Army Medical Center
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States